CLINICAL TRIAL: NCT06973603
Title: Exposure to Persistent Organic Pollutants and Severity of Endometriosis in the ComPaRe-Endometriosis Cohort
Acronym: POPENDO
Status: Not yet recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C24-04; ID-RCB (Other: 2025-A00414-45)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
Keywords: exposition; Endometriosis; Organic Persistent Polluant; Endometriosis severity; endomestriosis symptoms; endometriosis pain
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24mL blood sample (3 dry tubes with 8mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples — 24mL blood sample (3 dry tubes with 8mL)

SUMMARY:
Endometriosis is a chronic inflammatory disease affecting ~10% of women of childbearing age. It is characterized by the presence of endometrial-like tissue outside the uterus, causing lesions and adhesions between the organs, and is often accompanied by intense pain and sometimes infertility. The four-stage classification based on the severity of lesions does not always reflect the severity of symptoms. Adenomyosis, a similar pathology, is often present in the same patients, although it is now considered distinct from endometriosis. Diagnosis usually takes a long time, with an average delay of 7 years. The cause of the disease remains unknown, but hormonal, genetic and environmental factors, such as exposure to endocrine disruptors, are suspected. Persistent organic pollutants (POPs), such as dioxins and PCBs, may influence the risk and severity of the disease. Although experimental studies suggest a link between these substances and the progression of endometriosis, epidemiological research on the subject is still limited.

The central hypothesis of the POPENDO project is that higher concentrations of persistent organic pollutants (POPs) are associated with increased severity of endometriosis. The aim of the study is to explore the associations between serum levels of four families of POPs (PCBs, organochlorine pesticides, PFAS and BFR) and endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* ComPaRe participants ⩾ 18 years old. All ComPaRe participants are at least 18 years of age, so our research participants will all be adults.
* Having declared in ComPaRe that they had endometriosis
* Living in the Ile-de-France region (departments 75, 77, 78, 91, 92, 93, 94 or 95);
* Have given electronic consent stating: "By checking this box, I agree to be solicited for research outside ComPaRe"; This criterion is collected at the time of ComPaRe registration, when consent is collected. Participants can withdraw this consent at any time on their secure personal online account on the ComPaRe platform.
* Aged ≤ 45 years to avoid including premenopausal or menopausal women;
* In possession of MRI images used to diagnose their endometriosis (CD-ROM) that are no more than 5 years old;
* Enrolled in or benefiting from a social security scheme.

Exclusion Criteria:

* - People with contraindications to blood sampling will not be included in this research:
* Known severe anemia
* Hemophilia/coagulation disorders/anticoagulant use
* People with HIV, HBV or HCV will not be included in this study due to the risk of BSE (Blood Exposure Accident).
* Based on factors that may disrupt lipid dynamics and lipid pollutants, the following individuals will not be included:
* Pregnant and breast-feeding women
* People suffering from any of the following diseases:

  * Cancer
  * Morbid obesity (BMI>40)
  * Non-alcoholic steatohepatitis (NASH)
* Persons under court protection/guardianship/guardianship will not be able to participate in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be a group of female volunteers who have self-reported endometriosis. The group size will be a random sample of 650 women from the ~10,000 participants included in the ComPaRe-Endometriosis sub-cohort.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the severity of endometriosis, defined by the type of disease. | During 3 last years of analysis
  Analysis of several online questionnaires on endometriosis by participants
Evaluation of serum levels of polychlorinated biphenyls (PCBs) | 5 months after inclusion start until analysis of the last participant' blood sample
  Chemical analysis of participants' blood samples by the LABERCA laboratory
Evaluation of serum levels of per- and polyfluoroalkylates (PFAS) | 5 months after inclusion start until analysis of the last participant' blood sample
  Chemical analysis of participants' blood samples by the LABERCA laboratory
Evaluation of serum levels of Brominated flame retardants polluent (BFRs) | 5 months after inclusion start until analysis of the last participant' blood sample
  Chemical analysis of participants' blood samples by the LABERCA laboratory
Evaluation of serum levels of organochlorine pesticides (POCs) | 5 months after inclusion start until analysis of the last participant' blood sample
  Chemical analysis of participants' blood samples by the LABERCA laboratory

SECONDARY OUTCOMES:
definition of the level of severity of endometriosis by the rASRM stage (revised stage of the American Society for Reproductive Medicine) | During 3 last years of analysis
  Analysis of online questionnaires on endometriosis and rASRM stage
definition of the level of severity of endometriosis by the anatomical extension of the disease observed on MRI | During 3 last years of analysis
  Pelvic MRI images will be reviewed by radiologists from Hôpital Paris Saint Joseph to map endometriosis across 21 anatomical structures within 5 pelvic segments, using the ENZIAN classification to assess lesion location and severity.
endometriosis severity level defined by the severity of painful symptoms. | During 3 last years of analysis
  Analysis of annual follow-up questionnaire of ComPaRe-Endometriosis study participant assessing the severity of various pain types over the past three months using a numeric rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: MARINA Kvaskoff, Dr, Study Director — Hôpital Paul Brousse
Locations (1):
- Hôpital Paris Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided